CLINICAL TRIAL: NCT01906528
Title: The Pharmacodynamics of Mivacurium in Males and Females: A Study in Human Volunteers
Brief Title: Sex-related Differences in the Response to the Muscle Relaxant Drug Mivacurium
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB11-07970
Record Dates: First submitted 2013-07-17; First posted 2013-07-24 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: Muscle Relaxation; Sex
Keywords: Nondepolarizing neuromuscular blocking drug; Mivacurium; Sensitivity; Sex
MeSH Terms: conditions — Coitus; Hypersensitivity | interventions — Mivacurium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Males vs females (Experimental): Constant-rate IV infusions of Mivacurium, range 1.0 - 3 micro/kg/min, duration 150 - 180 min
  Interventions: Drug: Mivacurium

INTERVENTIONS:
Drug: Mivacurium — Effect of Mivacurium in males vs females
  Other Names: Mivacron

SUMMARY:
Muscle relaxants are drugs providing muscle relaxation during surgical treatment. Previous studies have shown that males and females respond differently to this kind of drug. Our hypothesis is that males are more sensitive to the effect of Mivacurium (a muscle relaxant) than females, meaning that males need a lower blood concentration of the drug than females in order to obtain a given effect.

DETAILED DESCRIPTION:
Muscle relaxants are a type of drug used to provide muscle relaxation during induction of anesthesia and surgical treatment. Residual drug effect postoperatively (i.e. residual muscle relaxation) occurs frequently and studies have shown that this may be harmful in certain groups of patients. Of special concern is residual effect on upper airway and breathing muscles. A previous study has shown that males and females respond differently to the effect of this kind of drug. It appears that some muscle groups which are important for airway protection and breathing are more sensitive to the effect of muscle relaxants in males than females. Males may therefore be more susceptible to postoperative lung complications than females. In this study we try to determine what causes the observed sex-related difference in response to the muscle relaxant Mivacurium. We have previously shown that this sex-related difference cannot be explained by different pharmacokinetics (what the body does to the drug) in males and females. Our hypothesis is that a pharmacodynamic (what the drug does to the body) difference between sexes exists, i.e. that a lower blood concentration of Mivacurium is needed in males than females in order to obtain a predefined degree of muscle relaxation in certain muscle groups.

ELIGIBILITY:
Inclusion Criteria: Healthy individuals with no current medication -

Exclusion Criteria: Previous complications during anesthesia, pregnancy, allergy to muscle relaxants, smoking, gastrointestinal reflux.

-

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2013-03; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics of Mivacurium | 6 months
  The mivacurium drug concentration in the blood associated with 50% of maximal drug effect at steady-state conditions (Css50) will be determined at the thumb and the handgrip muscles.

SECONDARY OUTCOMES:
Clearance of Mivacurium | 6 months
  Clearance calculated as the relationship between steady-state infusion rate of Mivacurium and Mivacurium blood concentration.

OTHER OUTCOMES:
Relationship between thumb acceleration (TOF ratio) and handgrip strength in both sexes | 6 months
  Thumb acceleration secondary to nerve stimulation at the ulnar nerve (TOF ratio) is an objective way of monitoring the effect of muscle relaxants that is used frequently during clinical anesthesia. Handgrip strength will be monitored with a dynamometer.

CONTACTS AND LOCATIONS:
Overall Officials: John R Feiner, MD, Principal Investigator — University of California, UCSF, San Francisco, USA
Locations (1):
- University of California, UCSF, San Francisco, California, United States